CLINICAL TRIAL: NCT01976273
Title: A Pilot Study Comparing the Efficacy of 1064 Q-switch Laser vs. Glycolic Acid Peels for the Treatment of Melasma: A Randomized Control Trial
Brief Title: A Pilot Study Testing 1064nm Q-switch Laser Versus Glycolic Acid Peels for the Treatment of Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU84150
Record Dates: First submitted 2013-10-15; First posted 2013-11-05 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Melanosis
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1064nm Q-switch Laser (Active Comparator): The 1064 Q-Switch Laser is a medical device that uses a focused laser to remove dark pigment (color) from the skin.
  Interventions: Device: 1064nm Q-switch Laser
- Glycolic Acid Peels (Active Comparator): A Glycolic Acid Chemical Peel is a mild skin treatment used to correct uneven texture and color by removing dead cells from the skin's outermost layer.
  Interventions: Other: Glycolic Acid Peels

INTERVENTIONS:
Device: 1064nm Q-switch Laser
  Arms: 1064nm Q-switch Laser
Other: Glycolic Acid Peels
  Arms: Glycolic Acid Peels

SUMMARY:
The purpose of this study is to find out the safety and effectiveness of 1064 Q-Switch Laser Therapy compared to Glycolic Acid Chemical Peels for the treatment of melasma.

DETAILED DESCRIPTION:
Participants in this study will be patients at the dermatology clinic who are clinically diagnosed with at least a 2X2 cm patch of melasma on each side of their face (forehead or cheek). Starting at 2 weeks before treatment (week 2), both sides will be pretreated and primed with 4% hydroquinone with, if necessary, 2.5% hydrocortisone cream BID. On the treatment day (2-weeks) and 6-weeks one half of the subject's face will receive glycolic acid peels and the other half of the face will receive 1064nm Q-switch laser. This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years or older
2. Subjects with at least a 2 x 2 cm patch of melasma on each side of the face (forehead or cheek)
3. Subjects in general good health
4. Subjects must be willing and able to understand and provide informed consent for the use of their tissue and communicate with the investigator
5. Subjects must be willing to not apply other treatment options for melasma during the course of the study

Exclusion Criteria:

1. Subjects under 18 years of age
2. Subjects who are pregnant and/or lactating
3. Subjects who are unable to understand the protocol or to give informed consent
4. Subjects diagnosed with mental illness
5. Subjects who have concurrent active uncontrolled disease to facial area (i.e uncontrolled acne)
6. Subjects who have had a chemical peel in the past 3 months
7. Subjects who have used a prescribed retinoid in the past 3 months
8. Subjects with a bleeding disorder
9. Subjects with a history of abnormal wound healing
10. Subjects with a history of abnormal scarring
11. Subjects who report being allergic to glycolic acid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01-07 (Actual); Study Completion 2015-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Q-switch Laser Left, Glycolic Acid Peels Comparator Right: The unit of randomization was the subject who was randomized 1:1 to receive glycolic acid peel on one side of the face, while the contralateral side of the face received the 1064nm Q-switch laser.
  Subjects in this arm were randomized to receive the interventions: 1064nm Q-switch laser on the left side of their face, and the glycolic acids peels on the right side of their face.
- Glycolic Acid Peels Comparator Left, Q-Switch Laser Right: The unit of randomization was the subject who was randomized 1:1 to receive glycolic acid peel on one side of the face, while the contralateral side of the face received the 1064nm Q-switch laser.
  Subjects in this arm were randomized to receive the interventions: 1064nm Q-switch laser on the right side of their face, and the glycolic acids peels on the left side of their face.
Period: Overall Study
Arm/Group | Q-switch Laser Left, Glycolic Acid Peels Comparator Right | Glycolic Acid Peels Comparator Left, Q-Switch Laser Right
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Q-switch Laser Left, Glycolic Acid Peels Comparator Right | Glycolic Acid Peels Comparator Left, Q-Switch Laser Right | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.78 (10.62) | 44.11 (11.94) | 42.94 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 8 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) of Improvement Rated by a Blinded Dermatologist From at Week 10
Description: The primary outcome was a blinded rating of improvement of the treatment area (1064nm Q-switch Laser Versus Glycolic Acid Peels) using a Visual Analog Scale (VAS). A dermatologist blindly evaluated the treated areas of each side from live subjects at baseline on the final follow up visit (week 10). The VAS of improvement was rated on a scale of 0 to10, with 0 being no improvement and 10 being the most improvement seen by the treatment.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 1064nm Q-switch Laser: The 1064 Q-Switch Laser is a medical device that uses a focused laser to remove dark pigment (color) from the skin.
  1064nm Q-switch Laser
- Glycolic Acid Peels: A Glycolic Acid Chemical Peel is a mild skin treatment used to correct uneven texture and color by removing dead cells from the skin's outermost layer.
  Glycolic Acid Peels
Arm/Group | 1064nm Q-switch Laser | Glycolic Acid Peels
Number analyzed (Participants) | 18 | 18
units on a scale | 4.37 (2.49) | 4.62 (3.41)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 1064nm Q-switch Laser | Glycolic Acid Peels
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1064nm Q-switch Laser (N=20) | Glycolic Acid Peels (N=20)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blistering/Scabbing (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes